CLINICAL TRIAL: NCT04965350
Title: A Phase III, Randomized, Double-blind Study to Assess the Consistency of the Immunogenicity of Three Consecutive Production Lots of Bivalent HPV Vaccine in Healthy Female Subjects Aged 9 - 30 Years and to Demonstrate Non-inferiority of the Candidate HPV Vaccine Manufactured at Commercial Scale Compared With a Pilot Scale
Brief Title: Lot Consistency Clinical Trial of Bivalent HPV Vaccine in 9 to 30 Years Old Healthy Females
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Collaborators: Yuxi Zerun Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 311-HPV-1005
Record Dates: First submitted 2021-06-21; First posted 2021-07-16 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2vHPV Consistency Lot 1 (Experimental)
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Pichia pastoris)
- 2vHPV Consistency Lot 2 (Experimental)
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Pichia pastoris)
- 2vHPV Consistency Lot 3 (Experimental)
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Pichia pastoris)
- 2vHPV Pilot Scale Lot (Active Comparator)
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Pichia pastoris)

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Pichia pastoris) — sterile solution for intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of three consecutive lots of bivalent HPV (Type 16,18) vaccine (Pichia pastoris) in healthy female subjects aged 9 - 30 years, and demonstrate the non-inferiority of the candidate HPV vaccine manufactured at commercial scale compared with a pilot scale.

ELIGIBILITY:
Inclusion Criteria:

* 9-30 healthy female able to provide legal identification.
* Written informed consent had to be obtained from the subject prior to enrolment (for subjects below the legal age of consent, written informed consent had to be obtained from a parent or legal guardian of the subject and, in addition, the subject had to sign and personally date a written informed assent).
* Women of child-bearing age(WOCBA): Subject had to have a negative urine pregnancy test, no plan to be pregnant in 7 months, and agree to use adequate contraceptive precautions during study period.

Exclusion Criteria:

* Subject has received a marketed HPV vaccine or participated in an HPV vaccine clinical trial.
* History of abnormal cervical screen test result (ASC-US or worse) or history of genital warts.
* History of severe allergic reaction that required medical intervention.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines.
* Pregnant or breastfeeding, or within 6 weeks after the end of pregnancy.
* Fever prior to vaccination (auxiliary temperature ≥37.3 °C).
* Hypertension (physical examination systolic blood pressure 140mmHg and or diastolic blood pressure 90mmHg.
* Received live attenuated vaccine within 15 days before vaccination or subunit or inactivated vaccine within 7 days.
* Received immunoglobulin and/or blood product 3 months prior to the first vaccination.
* Acute diseases or acute stage of the chronic diseases within 3 days preceding the vaccination.
* According to the judgment of the investigator, subject has or had any other symptoms, medical history and other factors that are not suitable for participating in this clinical trial.

Ages: 9 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 1100 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titers (GMTs) for HPV-16 and/or HPV-18 at one month post 3rd dose | At Month 7
Percentage of participants who seroconvert to HPV-16 and/or HPV-18 at one month post 3rd dose | At Month 7
  Seroconversion was defined as: For initially seronegative subjects [antibody titer below (<) 1:40 prior to vaccination], antibody titer greater than or equal to (≥) 1:40 after vaccination; For initially seropositive subjects (antibody titer ≥ 1:40 prior to vaccination), antibody titer after vaccination ≥ 4 fold the pre-vaccination antibody titer.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAE) during 30 days after each dose | 0~30 days after each vaccination
Incidence of solicited adverse events (AEs) after vaccination | 0~7 days after each vaccination
Incidence of unsolicited AEs after vaccination | 0~30 days after each vaccination
Incidence of serious adverse events (SAEs) | Month 0 to Month 7

CONTACTS AND LOCATIONS:
Overall Officials: Ting Huang, Principal Investigator — Sichuan Center for Disease Control and Prevention
Locations (1):
- Mianyang Center for Disease Control and Prevention, Mianyang, Sichuan, China